CLINICAL TRIAL: NCT01268566
Title: A Phase 2 Study of MEDI-575 in Adult Subjects With Recurrent Glioblastoma Multiforme
Brief Title: A Study of MEDI-575 in Subjects With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI-575-1042
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Tovetumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDI-575, 25 mg/kg (Experimental): MEDI-575 administered as an intravenous infusion at 25 mg/kg over a period of 60-minutes on Day 1 of each 21-day cycle until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, or other reasons for participants withdrawal.
  Interventions: Drug: MEDI-575

INTERVENTIONS:
Drug: MEDI-575 — MEDI-575 as an IV infusion.

SUMMARY:
The primary objective of this Phase II study is to evaluate the progression-free survival at 6 months in adult subjects with a first recurrence of Glioblastoma Multiforme who are treated with MEDI-575.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open-label, single-arm study to evaluate the antitumor activity, safety, and pharmacology of MEDI-575 in adult subjects with first recurrence of GBM.

Approximately 55 subjects will be enrolled to determine the preliminary efficacy profile of MEDI-575 in the treatment of subjects with first recurrence of GBM. Subjects will receive MEDI-575 as a 60-minute IV infusion on Day 1 every 21 days until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, or other reasons for subject withdrawal.

The primary assessment of antitumor activity is PFS-6; tumor response and progression will be determined using Updated Response Assessment Criteria of High Grade Gliomas- Neuro-Oncology Working Group v.1. Approximately 15 investigational sites in the United States will participate in this study. All subjects will be followed every 3 months for the duration of the trial (defined as 9 months from the date the last subject is entered into the trial or when the sponsor stops the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization (applies to covered entities in the USA only) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Age ≥18 years old at the time of screening
* Histologically confirmed diagnosis of World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma)
* Previous first line treatment with radiotherapy and temozolomide (treatment prior to radiation and temozolomide permitted, [ie, Gliadel])
* Documented first recurrence of GBM by diagnostic biopsy or by contrast-enhanced magnetic resonance imaging (MRI) as per Updated Response Assessment Criteria of High Grade Gliomas- Neuro-Oncology Working Group (Wen et al, 2010)
* Life expectancy ≥ 12 weeks
* Adequate hematologic and organ function
* Negative serum pregnancy test (women only)
* Two methods of birth control for female participants of child-bearing potential or male participants with their female partners of child-bearing potential

Exclusion Criteria:

* Treatment with any chemotherapy, radiotherapy, immunotherapy, biologic, hormonal therapy or investigational agent 30 days prior to study entry
* Concurrent enrollment in another clinical study involving an investigational agent
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals
* Previous mAb treatment specifically directed against PDGF or PDGF receptors
* Previous bevacizumab or other VEGF and anti-angiogenic treatment
* More than 1 recurrence of GBM
* Any surgery (not including minor diagnostic procedures) within 2 weeks prior to baseline disease assessments; or not fully recovered from any side effects of previous procedures
* History of serious allergy or reaction to any component of the MEDI-575 formulation
* New York Heart Association ≥ Grade 2 congestive heart failure within 6 months prior to study entry
* Uncontrolled or significant cardiovascular disease
* History of other invasive malignancy within 5 years prior to study entry except for cervical carcinoma in situ (CIS), non-melanomatous carcinoma of the skin or ductal carcinoma in situ (DCIS) of the breast that have been surgically cured
* History of active human immunodeficiency virus or active hepatitis B or C viral infection will be excluded to eliminate the risk of increased AEs due to immune compromise.
* Systemic immunosuppressive therapy.
* Subjects taking corticosteroids must be on a stable dose for 7 days prior to initiation of treatment with MEDI-575 16) Presence of extracranial metastatic or leptomeningeal disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Stanford, California
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Canton, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Seattle, Washington

REFERENCES:
- See also: CD-ON-MEDI-575-1042 Redacted CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=5&filename=1042%20Protocol%20V%202%2019-May-11_Redacted-IP%20Comments.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 subjects were enrolled and treated at 13 sites in the United States.
Pre-assignment Details: A total of 62 participants were screened. Of which, 56 participants were enrolled into study as 5 participants failed screening and 1 participant withdrew consent.
Groups:
- MEDI-575, 25 mg/kg: MEDI-575 administered as an intravenous infusion at 25 mg/kg over a period of 60-minute on Day 1 of each 21-day cycle until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, or other reasons for participant withdrawal.
Period: Overall Study
Arm/Group | MEDI-575, 25 mg/kg
Started | 56
Completed | 13
Not Completed | 43
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 12
Not completed — Death | 30

BASELINE CHARACTERISTICS:
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 6 Months
Description: Progression-free survival (PFS) rate at 6 months is defined as the proportion of participants who neither progressed nor died before 6 months after the first dose. Progression was determined using Updated Response Assessment Criteria of High Grade Gliomas: Response Assessment in Neuro-Oncology Working Group (RANO criteria). Progression was defined as at least 25% increase in measurement of enhancing lesions compared with the smallest tumor measurement obtained during the study; or significant increase in T2/fluid attenuated inversion recovery (FLAIR) nonenhancing lesion compared with baseline scan or best response; or any new lesion; or clear clinical deterioration; or failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease. PFS-6 was estimated using Kaplan-Meier method.
Time Frame: 6 months
Population: Intent-to treat (ITT) population: All participants who entered into the study (ie, participants for whom investigator notified the interactive web response system [IWRS] that the participant met eligibility criteria and the IWRS assigned unblinded study drug to the participant).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Percentage of participants | 15.4 [8.1 to 24.9]

2. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response rate is calculated based upon the disease assessments recorded during the study visits using RANO criteria. Best overall response includes complete response (CR), CR with confirmation, partial response (PR), PR with confirmation, stable disease and progressive disease. Confirmed responses are those that persist on repeat imaging studies at least 4 weeks after the initial documentation of response.
Time Frame: Study entry through the end of the study, up to 21 months
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Percentage of participants
  Complete response with confirmation | 0
  Complete response without confirmation | 0
  Partial response with confirmation | 0
  Partial response without confirmation | 0
  Stable disease | 41.1
  Progressive disease | 55.4
  Unknown | 3.6

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate (ORR) is defined as the proportion of participants with confirmed CR or confirmed PR using RANO criteria. Confirmed CR and PR are those that persist on repeat imaging study for at least 4 weeks after the initial documentation of the response. CR is defined as complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks, no new lesions, stable or improved nonenhancing (T2/FLAIR) lesions, patient is off corticosteroids and stable or improved clinically. PR is defined as 50% decrease compared with baseline in the measurement of all measurable enhancing lesions sustained for at least 4 weeks, no progression of nonmeasurable disease, no new lesions, stable or improved nonenhancing (T2/FLAIR) lesions, no increase in the corticosteroid dose and stable or improved clinically.
Time Frame: Study entry through the end of the study, up to 21 months
Population: ITT population
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Percentage of participants | 0 [0.0 to 5.2]

4. Secondary Outcome: Time to Response
Description: Time to response (TTR) is defined as the time from the study entry to the first documentation of confirmed CR or confirmed PR. Analysis was based on responses confirmed at a repeat assessment made at least 4 weeks after the initial response, with the TTR taken as the first time the response was observed, not the confirmation assessment. TTR was estimated using Kaplan-Meier method.
Population: ITT population with an objective response (ie, confirmed CR or PR) were assessed. TTR was not estimable as there were no participants with an objective response.
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the duration from the first documentation of objective disease response (ie, confirmed CR or confirmed PR) to the first documented disease progression. Duration of response was estimated using Kaplan-Meier method and evaluated only for the participants of subgroup with an objective response.
Population: ITT population with an objective response (ie, confirmed CR or PR) were assessed. Duration of response was not estimable as there were no participants with an objective response.
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is defined as time from the start of treatment with MEDI-575 until the documentation of disease progression. Disease progression was defined by at least 25% increase in measurement of enhancing lesions compared with the smallest tumor measurement obtained during the study; or significant increase in T2/FLAIR nonenhancing lesion compared with baseline scan or best response; or any new lesion; or clear clinical deterioration; or failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease. TTP was estimated using Kaplan-Meier method.
Time Frame: Study entry until the first documented disease progression, up to 16 months
Population: ITT population. N= number of participants analyzed for this outcome measure
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 48
Months | 1.4 [1.4 to 1.8]

7. Secondary Outcome: Progression-free Survival Rate at 3 Months and 9 Months
Description: PFS rate at 3 and 9 months is defined as proportion of participants who neither progressed nor died due to any cause, whichever occurred first after first dose at 3 months and 9 months, respectively. Progression was defined as at least 25% increase in measurement of enhancing lesions compared with the smallest tumor measurement obtained during the study; or significant increase in T2/FLAIR nonenhancing lesion compared with baseline scan or best response; or any new lesion; or clear clinical deterioration; or failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease. Proportion of participants with PFS at 3 and 9 months were estimated using Kaplan-Meier method.
Time Frame: 3 months and 9 months
Population: ITT population
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Percentage of participants
  PFS rate at 3 months | 26.5 [17.1 to 36.7]
  PFS rate at 9 months | 8.8 [3.6 to 17.1]

8. Secondary Outcome: Progression-free Survival
Description: PFS was measured from the start of treatment with MEDI-575 until the documentation of disease progression or death due to any cause, whichever occurred first. Progression was defined as at least 25% increase in measurement of enhancing lesions compared with the smallest tumor measurement obtained during the study; or significant increase in T2/FLAIR nonenhancing lesion compared with baseline scan or best response; or any new lesion; or clear clinical deterioration; or failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease. PFS was censored on the date of last tumor assessment documenting absence of tumor progression for participants who have no documented progression and were still alive prior to data cutoff, dropout, or the initiation of alternate anticancer treatment. Time to PFS was estimated using Kaplan-Meier method.
Time Frame: 9 months
Population: ITT population. N= number of participants analyzed for this outcome measure
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 50
Months | 1.4 [1.4 to 1.8]

9. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the start of treatment with MEDI-575 until death. For the participants who were alive at the end of study or lost to follow-up, Overall survival was censored on the last date when participants were known to be alive. The Overall survival was estimated using the Kaplan-Meier method.
Time Frame: Study entry to death, up to 16 months
Population: ITT population. N= number of participants analyzed for this outcome measure
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 30
Months | 9.7 [6.5 to 11.8]

10. Secondary Outcome: Percentage of Participants With Expression of PDGFR Alpha in the Tumor Samples
Description: MEDI-575 (study drug) blocks platelet-derived growth factor (PDGF) binding to PDGF receptor (PDGFR) alpha and inhibits signaling. The tissue samples which were collected prior to the study entry (archived tumor samples) were evaluated by immunohistochemistry staining for expression of PDGFR alpha signaling protein that are targets of MEDI-575. Expression of PDGFR alpha in tumor cells and tumor-associated stromal cells were evaluated for intensity and distribution of staining. The percentage of participants with positive PDGFR alpha staining in the tumor cells and tumor-associated stromal cells were reported.
Time Frame: Screening (Day-28 to Day -1)
Population: ITT population with archived tumor samples were assessed.
Measure: Number; unit: Percentage of participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 39
Percentage of participants
  Positive PDGFR alpha staining in tumor cells | 46
  Positive staining in tumor stromal cells | 26

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Treatment-emergent AEs (TEAEs) are AEs occurring or worsening after the administration of study drug until 90 days after the last dose of study drug or until the participant began another anticancer therapy, which ever came first. A serious AE (SAE) is any AE that results in death, is immediately life threatening, require (or prolong) inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above. The TEAEs and SAEs were summarized using MedDRA version 15.1. Participants were counted only once for each event, regardless of number of events the participant had.
Time Frame: Baseline to last record on study, up to 21 months
Population: Safety population included all participants who received at least 1 dose of MEDI-575.
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Participants
  Participants with TEAEs | 50
  Participants with treatment emergent SAEs | 17

12. Secondary Outcome: Number of Participants With Worst ECOG Performance Status On-study and Last Record On-study
Description: Eastern Cooperative Oncology Group (ECOG) performance status is a scale that measures how cancer affects the daily life of a participant on an ordinal scale from grade 0 (fully active ie, best) to 5 (dead ie, worst). Following are ECOG grades: 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair. 5: Dead.
Time Frame: Baseline to last record on study, up to 21 months
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Participants
  Worst on-study: Grade 0 | 6
  Worst on-study: Grade 1 | 24
  Worst on-study: Grade 2 | 16
  Worst on-study: Grade 3 | 9
  Worst on-study: Grade 4 | 1
  Worst on-study: Not done | 0
  Last record on-study: Grade 0 | 9
  Last record on-study: Grade 1 | 27
  Last record on-study: Grade 2 | 12
  Last record on-study: Grade 3 | 7
  Last record on-study: Grade 4 | 1
  Last record on-study: Not done | 0

13. Secondary Outcome: Treatment-emergent Adverse Events Related to Laboratory Parameters
Description: Laboratory evaluations of blood and urine samples were performed, including hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count with differential); serum chemistry (calcium, chloride, magnesium, potassium, sodium, aspartate transaminase, alanine transaminase, alkaline phosphatase, gamma glutamyl transferase, lactic dehydrogenase, carbon dioxide/bicarbonate, blood urea nitrogen, uric acid, creatinine, total bilirubin, glucose, albumin, total protein, triglycerides, cholesterol, phosphorous); urinalysis (pH, protein, blood, glucose, ketones, bilirubin); and coagulation parameters. Abnormal laboratory finding that required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation, was reported as an AE. Number of participants with TEAEs related to laboratory evaluations were reported.
Time Frame: Baseline to last record on study, up to 21 months
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Participants
  Anaemia | 1
  Thrombocytopenia | 2
  Activated partial thromboplastin time prolonged | 1
  Lymphocyte count decreased | 1
  Platelet count decreased | 1
  White blood cell count increased | 1
  Blood lactate dehydrogenase increased | 1
  Hypokalaemia | 1
  Hypomagnesaemia | 1
  Hypophosphataemia | 1
  Haematuria | 2
  Urinary tract infection | 4

14. Secondary Outcome: Treatment-emergent Adverse Events Related to Electrocardiogram Evaluations
Description: All 12-lead electrocardiograms (ECGs) performed during the study were obtained in triplicate (ie, 3 ECGs were obtained within a 5-minute time period) and analyzed. Number of participants with TEAEs related to ECG after the start of study drug administration were reported. Participants were counted only once for each system organ class and preferred term, regardless of how many events the participants had.
Time Frame: Baseline to last record on study, up to 21 months
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Participants
  Abnormal ECG T wave | 1
  Bradycardia | 1
  Sinus bradycardia | 1

15. Secondary Outcome: Treatment-emergent Adverse Events Related to Vital Sign Parameters
Description: Vital sign assessments were conducted throughout the study and included body temperature, blood pressure (seated), pulse rate and respiratory rate. The TEAEs related to vital signs in participants were reported. Participants were counted only once for each system organ class and preferred term, regardless of how many events the participants had.
Time Frame: Baseline to last record on study, up to 21 months
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | MEDI-575, 25 mg/kg
Number analyzed (Participants) | 56
Participants
  Hypertension | 2
  Hypotension | 2
  Heart rate increased | 1
  Pyrexia | 1

ADVERSE EVENTS:
Time Frame: Baseline to last record on study, up to 21 months
Arm/Group | MEDI-575, 25 mg/kg
Serious Adverse Events (participants affected / at risk) | 17/56
Other Adverse Events (participants affected / at risk) | 43/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-575, 25 mg/kg (N=56)
Cardiac failure (Cardiac disorders) | 1 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Cerebral cyst (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (4)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI-575, 25 mg/kg (N=56)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 13 (18)
Nausea (Gastrointestinal disorders) | 13 (16)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 16 (19)
Gait disturbance (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 5 (5)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (6)
Aphasia (Nervous system disorders) | 7 (9)
Cognitive disorder (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 7 (8)
Headache (Nervous system disorders) | 9 (11)
Hemiparesis (Nervous system disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 6 (6)
Confusional state (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.